CLINICAL TRIAL: NCT06211699
Title: The Effect of Omentopexy and Clips on the Staple Line During Laparoscopic Sleeve Gastrectomy on Early Postoperative Outcomes: A Randomized Trial
Brief Title: Effect of Clips Versus Omentopexy on Postoperative Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdullah Sisik, Associate Prof., FEBS-MIS, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 218494864
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Bleeding; Postoperative Complications; Postoperative Nausea and Vomiting
Keywords: Laparoscopic Sleeve Gastrectomy; Bleeding; Staple Line Reinforcement; Postoperative First Month Readmission
MeSH Terms: conditions — Hemorrhage; Postoperative Complications; Postoperative Nausea and Vomiting | interventions — Surgical Instruments

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The primary surgeon is naturally not blinded to the patient groups and the other surgeon who records and evaluates the data is blinded to the patient groups. The patient was blind to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omentopexy with Laparoscopic Sleeve Gastrectomy (Active Comparator): Patients who underwent continuous through-and-through omentopexy of the omentum to the remnant stomach staple line after resection during Laparoscopic Sleeve Gastrectomy (omentopexy group).
  Interventions: Procedure: Omentopexy with Laparoscopic Sleeve Gastrectomy
- Clips with Laparoscopic Sleeve Gastrectomy (Active Comparator): Patients who underwent consecutive clippping along the staple line of the remnant stomach during Laparoscopic Sleeve Gastrectomy (clips group)
  Interventions: Procedure: Clips with Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Omentopexy with Laparoscopic Sleeve Gastrectomy — Patients with omentum sewed to the remnant gastric staple line during laparoscopic sleeve gastrectomy.
  Arms: Omentopexy with Laparoscopic Sleeve Gastrectomy
Procedure: Clips with Laparoscopic Sleeve Gastrectomy — Patients performed clips to the remnant gastric staple line during laparoscopic sleeve gastrectomy
  Arms: Clips with Laparoscopic Sleeve Gastrectomy

SUMMARY:
In this prospective randomized study, patients were divided into two groups: clips group and omentopexy group. The groups were compared in terms of postoperative decrease in hemoglobin and hematocrit values, preoperative and peroperative blood pressure values, duration of surgery, number of patients requiring erythrocyte suspension (ES) transfusion, length of hospital stay, hospital readmissions in the first 30-days postoperatively and early postoperative complications.

DETAILED DESCRIPTION:
This prospective randomized controlled trial was conducted at the University of Health Science Umraniye Training and Research hospital between July 2023 and November 2023. The Patients who underwent LSG, were between the ages of 18 and 65, with a Body Mass Index (BMI) ≥ 40 or BMI ≥ 35 with at least one obesity-related comorbidity were included in the study. Patients who underwent other bariatric surgery procedures, had uncontrolled hypertension, and had preoperative history of gastroesophageal reflux disease (GERD) symptoms were excluded. Approval for the study was received from the ethics committee of tertiary health institution (21.06.2023/218494864). Before the surgery, each of the participants were received comprehensive information about the study, the techniques to be applied were explained, they would be randomly assigned in one of the two groups and the consent form obtained in this context.

Study Groups In the study, patients were divided into two groups: Patients who underwent consecutive clippping along the staple line of the remnant stomach during LSG (clips group) and patients who underwent continuous through-and-through omentopexy of the omentum to the remnant stomach staple line after resection during LSG (omentopexy group).

Data Collection Age, gender, comorbidities, smoking history, preoperative height-weight-BMI values, preoperative systolic blood pressure (SBP)-diastolic blood pressure (DBP) values, preoperative hemoglobin-hematocrit values, peroperative SBP-DBP-mean blood pressure (MBP), duration of surgery, postoperative 6th hour and time of discharge hemoglobin-hematocrit values, number of patients transfused erythrocyte suspension (ES) or requiring invasive intervention due to bleeding, length of hospital stay, hospital readmissions in the first postoperative month, and early postoperative complications were recorded. Duration of surgery was determined from the first skin incision to the last skin suture.

Preoperative, peroperative and Postoperative Evaluation Preoperative anesthesia, cardiology and pulmonology evaluations were performed for each patient. Hepatobiliary ultrasound and upper gastrointestinal endoscopy evaluation were performed. Each patient was administered low molecular weight heparin (enoxaparin 6000 units 1x1 subcutaneously) 12 hours before surgery and was taken to surgery with antiembolism stockings. Intermittant pneumatic compressor device was used perioperatively. Omentopexy was performed with 3-0 V-loc suture (26 mm, V-20 Tapper) and clippping was performed with endo clips II (10 mm, medium/large). Since ERAS protocol was applied in our clinic, no drain was placed in any patient.

At the 4th postoperative hour, all patients were mobilized, intensive respiratory exercise was performed and clear liquid food was started. Complete blood count and C-reactive protein (CRP) laboratory parameters were checked at postoperative 6th, 24th and 48th hour (discharge). Vital parameters were checked every 6 hours postoperatively. Patients who have an acute decrease in hemoglobin value together with a pulse rate of 100 or more per minute and systolic/diastolic blood pressure values below 90/60 mmHg were considered as bleeding and erythrocyte suspension was transfused. Early on the second postoperative day, the patient who could tolerate oral food and did not require additional intervention was discharged.

The primary outcome of the study was to compare the two methods in terms of early postoperative bleeding. The seconder outcome of the study is to compare the groups in terms of duration of surgery, lengh of hospital stay and hospital readmission in the first 30-days postoperatively.

Randomization Patients were numbered according to the order of enrollment and randomly assigned 1:1 to the clips group or the omentopexy group. Allocations were generated using randomly permuted blocks (available at www.randomization.com). All randomization was done by an individual who wasn't included in the study, and the allocations were preserved in sealed envelopes. A research assistant opened the sealed envelope at the beginning of surgery, disclosing the patient's allocation group to the surgeon. The primary surgeon is naturally not blinded to the patient groups and the other surgeon who records and evaluates the data is blinded to the patient groups. All operations were performed laparoscopically by the same surgeon. Since this was a pilot study, no sample size was calculated.

Comparison of Groups The groups were compared in terms of postoperative decrease in hemoglobin and hematocrit values, preoperative and peroperative blood pressure values, duration of surgery, length of hospital stay, hospital readmissions in the first 30-days postoperatively, early postoperative complications and number of patients requiring ES transfusion.

Statical Analaysis A meticulous statistical evaluation was performed on the collected baseline clinical data to ensure robust and reliable conclusions. For continuous variables, the analysis employed both t-tests and Mann-Whitney U tests, depending on the distribution characteristics of the data. Categorical variables, on the other hand, were rigorously examined using either Fisher's exact test or the chi-square test, based on the appropriateness for the dataset at hand.

This analytical process was facilitated by the use of SPSS software, version 22.0 (IBM Corp., Armonk, NY), which is renowned for its precision and versatility in handling diverse statistical tasks. Care was taken to conduct all tests as two-tailed, providing a comprehensive view of the data. The threshold for statistical significance was set at a p value of less than 0.05, aligning with standard practices in clinical research.

ELIGIBILITY:
Inclusion Criteria:

* The Patients who underwent LSG
* Between the ages of 18 and 65,
* A Body Mass Index (BMI) ≥ 40 or BMI ≥ 35 with at least one obesity-related comorbidity

Exclusion Criteria:

* Patients who underwent other bariatric surgery procedures,
* Patients who declined to be participate
* uncontrolled hypertension
* preoperative history of gastroesophageal reflux disease (GERD) symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Postoperative Bleeding | up to 3 Months
  The primary outcome of the study was to compare the two methods in terms of early postoperative bleeding. This comparison will be made with hemoglobin and hematocrit values measured at postoperative 6th hour, 24th hour and at discharge. The groups will be compared according to the decrease in hemoglobin and hematocrit values, whether ES displacement is required, and whether intervention is required.

SECONDARY OUTCOMES:
Postoperative First Month Readmission | 30-days postoperatively
  The seconder outcome of the study is to compare the groups in terms of hospital readmission in the first 30-days postoperatively. Patients readmitted to the hospital in the first postoperative month will be recorded and reasons for readmission will be categorized and groups will be compared.
The duration of surgery (minutes) | Intraoperative
  The seconder outcome of the study is to compare the groups in terms of duration of surgery (minutes) Surgical time will be calculated based on the time between the first port incision and the last skin suture.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Taha Demirpolat, M.D., Study Director — Umraniye Education and Research Hospital
Locations (1):
- Umraniye Training and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No